CLINICAL TRIAL: NCT06366828
Title: Prediction Models for Complications After CRT in Esophageal Cancer
Acronym: MODELS
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other); Dutch Institute for Clinical Auditing (DICA) (Unknown); ZorgTTP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11446
Record Dates: First submitted 2024-02-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: The Aim of This Project is to Develop and Validate NTCP-models for Complications After nCRT (and Surgical Resection)
Keywords: prediction models; esophageal cancer (EC)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective — follow up

SUMMARY:
The aim of this project is to develop and validate NTCP-models for complications after nCRT (and surgical resection), that can be uses for model-based dose optimization for PhRT and PRT, and for model-based selection for PRT, in patients with esophageal cancer

DETAILED DESCRIPTION:
Plan of investigation

In the present project we aim to evaluate two potential strategies to predict and consider a broad spectrum of complications for radiotherapy plan optimization and patient selection:

A comprehensive set of separate NTCP-models for several cardiopulmonary and post-operative complications after nCRT, which results in an NTCP-profile.

A single multivariable NTCP-model for a so-called Complication Sum Score (CSS), which is a single composite complication endpoint including all complications after nCRT, weighted depending on severity and impact.

These prediction models can be used for RT plan optimization and patient selection.

In order to develop these prediction models the project consortium brings together existing prospective data registries for esophageal cancer, namely the Dutch Upper GI Cancer Audit (DUCA) and the Dutch Cancer Registry (NKR) (as well as the POCOP study).

The data of these registries will be linked to a retrospective radiotherapy database using the ProTRAIT infrastructure, resulting in a dataset of over 2000 patients.

In this retrospective cohort study, we will focus on esophageal cancer patients who were treated with nCRT, and for whom an esophagectomy was intended. We will include the patients who received nCRT and the esophagectomy in one of the participating centers. Patients who only received nCRT in one of the participating centers and for whom surgical resection was omitted will be included as well. Detailed eligibility criteria can be found in that section.

Eligible patients will be identified by the Dutch Cancer Registry. The surviving patients will be asked to provide informed consent for participation in this study, permission to combine the different data registries and for future use of their data. Patients who died will be included as well, unless they objected agains the use of there data in the participating centers.

Of the participating patients, the radiotherapy plan-CT and treatment plans (i.e. RTplan, RT struct, RT dose), will be pseudo-anonymized, uploaded and transferred to the UMCG data platform, by the participating radiotherapy centers.

A third trusted party, Zorg TTP, will be responsible for the pseudonymization of the three data sources; the Dutch upper GI cancer audit (DUCA), the Dutch Cancer Registry (NKR) and the RTregistry. After that the linkage will be performed at the UMCG.

ELIGIBILITY:
Inclusion Criteria:

* Tumor in the esophagus, histologically proven or suspect for esophageal carcinoma
* WHO performance 0-2
* Age>18years
* No distant metastasis (M0)
* Treated with nCRT and planned for or followed by an esophagectomy between 2015 and 2021 in one of the participating centers.

Exclusion Criteria:

* Sarcoma, neuro-endocrine or small cell carcinoma of the esophagus
* Patients who underwent a surgical resection in a non-participating surgical center will be excluded

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer, treated with nCRT between 2015-2021 in the participating centers. See eligibility criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Multivariable NTCP models will be developed for the prediction of the following | Within 90 days after surgery
  Postoperative complications (graded by ECCG classification (3) ):
  Atrial fibrillation ≥grade 2
  Pneumonia ≥grade 2
  Respiratory failure requiring re-intubation
  Anastomotic leakage ≥ grade 2
Cardiac events grade II or higher (CTCAE v 5.0), including: | 1 and 2 year after nCRT
  Pericardial effusion
  Myocardial infarction and other acute coronary events
  Heart failure Pericardial effusion
  Myocardial infarction and other acute coronary events
  Heart failure
  Atrial fibrillation
Mortality | 1 and 2 year after nCRT
  Mortality
Complication Sum Score, that will be determined in Delphi consensus | 1 year after nCRT
  Complication Sum Score, that will be determined in Delphi consensus

SECONDARY OUTCOMES:
Patient-rated dysphagia | Up to 30 days after nCRT
  Patient-rated dysphagia
Patient-rated nausea | Up to 30 day after nCRT
  Patient-rated nausea
Patient-rated fatigue / daily functioning | Up to 6 months after nCRT
  Patient-rated fatigue / daily functioning
Hospitalization after esophagectomy (days) | Hospitalization after esophagectomy, average 12 days
  Hospitalization after esophagectomy (days)
Intensive care unit stay after esophagectomy (days) | Intensive care unit stay after esophagectomy, average 1.5 days
  Intensive care unit stay after esophagectomy (days)

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastro clinic, Maastricht, Limburg
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Holland PTC, Delft
  - UMCG, Groningen
  - Zuyderland hospital, Heerlen
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided